CLINICAL TRIAL: NCT05707312
Title: Staging Endometrial caNcer Based on molEcular ClAssification
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: SENECA
Record Dates: First submitted 2023-01-18; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Endometrial Cancer; Lymph Node Metastasis; Sentinel Lymph Node
MeSH Terms: conditions — Endometrial Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- POLEmut (POLE mutant endometrial cancer patients): POLE mutant endometrial cancer patients
- MMRd (mismatch repair deficient endometrial cancer patients): mismatch repair deficient endometrial cancer patients
- NSMP (no specific molecular profile endometrial cancer patients to NSMP): no specific molecular profile endometrial cancer patients to NSMP
- p53abn (p53 abnormal endometrial cancer patients): p53 abnormal endometrial cancer patients

SUMMARY:
The SENECA study tries to evaluate the rate of lymph node involvement depending on the molecular subgroup in early-stage endometrial cancer (I/II) patients undergoing surgery as part of their treatment.

DETAILED DESCRIPTION:
The management of endometrial cancer (EC) is currently undergoing a true revolution in terms of diagnosis and treatment. Since 2013 and thanks to the TCGA project1 (The Cancer Genome Atlas), four distinct molecular subgroups (POLE, MMR-D, Copy number low, Copy number high) with distinct prognostic implications were identified.

Subsequently, PROMISE study2 brought this "new era" closer to daily clinical practice. These new findings led ESGO3 (European Society of Gynecologic Oncology) to decide to integrate this molecular classification into the definition of the different risk groups.

Currently, thanks to the retrospective analysis of the PORTEC-3 cohort4,5, we know that these four molecular subgroups may present differences in survival in high-risk patients depending on the type of treatment proposed, chemoradiotherapy vs. adjuvant radiotherapy. This question will be answered by the RAINBO trial6 (Refining Adjuvant treatment IN endometrial cancer Based On molecular profile).

On the other hand, the surgical management of early endometrial cancer (stage I/II) has been changing for some years now, especially with regard to nodal staging, from modulation of treatment depending on the risk group (pelvic lymphadenectomy +/- sentinel lymph node (SLN) for low and intermediate risk groups vs. aortopelvic lymphadenectomy +/- SLN for those at high risk) to a generalization of treatment based on detailed study of the sentinel node following the algorithm described by the group of Abu-Rustum NR et al7.

Just as the RAINBO study will try to clarify the type of adjuvant treatment necessary for each molecular subgroup, we do not currently know if it could be possible to tailor the type of lymph node staging in early EC (the most common and most frequent in our daily clinical practice) depending on the molecular subgroup8,9.

We therefore propose a study to evaluate the lymph node involvement rate depending on the molecular subgroup in early-stage EC (I/II).

ELIGIBILITY:
Inclusion Criteria:

* Patient was operated during 2021-2022
* Histological confirmation of Endometrial Cancer with endometrioid histology or high risk histology (serous, clear cell, carcinosarcoma and mixed histologies)
* Preoperative FIGO stage I or II by MRI or US
* Preoperative CT-Scan or PET-CT without evidence of local or distant disease (could be omitted in low-risk and intermediate risk endometrial carcinoma with low grade histology)
* Surgical protocol according to ESGO/ESTRO/ESP guidelines
* A detailed sentinel lymph node study protocol must be accredited, either by ultra-staging or OSNA
* Molecular analysis performed on the pathology specimen according to ESGO/ESTRO/ESP guidelines (POLE mutation analysis could be omitted in low-risk and intermediate risk endometrial carcinoma with low grade histology).

Exclusion Criteria:

* Pregnant women
* Previous hysterectomy
* Previous pelvic/para-aortic lymphadenectomy
* Presence of extra-uterine disease (peritoneal, visceral or suspicious lymph node metastasis)
* Past medical history of any invasive tumor
* History of previous abdominal or pelvic radiotherapy of any type (including braquitherapy)
* History of preoperative neoadjuvant chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with early-stage (FIGO stage I-II) EC that underwent surgical treatment with lymph node evaluation between January 2021 to December 2022, both included.
Sampling Method: Non-Probability Sample
Enrollment: 1032 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sentinel lymph node involvement rate | 1 month after the intervention/procedure/surgery
  Lymph node involvement rate (sentinel) for each molecular subtype in patients with stage I/II EC.(percentage)

SECONDARY OUTCOMES:
Lymph node involvement rate | 1 month after the intervention/procedure/surgery
  Lymph node involvement rate (sentinel and non-sentinel) for each prognostic risk group in patients with stage I/II EC.
Compliance of ESGO quality Indicators. | 1 month after the intervention/procedure/surgery
  Compliance of ESGO quality Indicators for center (percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Chiva, MD PHD, Principal Investigator — Clinica Universidad de Navarra
Locations (1):
- Clinica Universidad de Navarra, Pamplona, Navarre, Spain

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT05707312/Prot_SAP_000.pdf